CLINICAL TRIAL: NCT03744598
Title: An Observational Study of Self-monitoring of Spirometry and Symptoms Via the patientMpower App in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Self-monitoring of Spirometry & Symptoms Via patientMpower App in Idiopathic Pulmonary Fibrosis
Status: Terminated | Type: Observational
Why Stopped: Clinic visits stopped due to COVID19
Sponsor: patientMpower Ltd. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: IPF patientMpower 03
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single-arm, open-label observational study in idiopathic pulmonary fibrosis (IPF) patients receiving usual care at an interstitial lung disease specialist center. The objectives are [1] to characterise the longitudinal trends of patient-measured Forced Vital Capacity (FVC) and impact of IPF on daily life Patient Reported Outcome Measures (PROM) in a cohort of patients with IPF [2] to determine the correlation (if any) between patient-measured FVC and PROMs with clinic-observed measurements and [3] to assess if longitudinal trends in patient-measured FVC are predictive of clinical health outcomes in IPF. An additional purpose is to assess the acceptability and utility of the patientMpower app in helping IPF patients and their healthcare professional caregivers manage their condition. Patients will record FVC, symptoms (e.g. dyspnea) and activity (step count) daily and PROM once a week on the patientMpower app.

The planned observation period is sixteen weeks. No additional clinic visits are required (versus usual care). In-clinic assessments of lung function, dyspnea and PROM will be done at baseline and study end. Patients and healthcare professionals will provide their opinion on utility and acceptability of patientMpower app at study end.

DETAILED DESCRIPTION:
This is a single-arm, open-label observational study in IPF patients receiving usual care at an interstitial lung disease specialist centre. The objectives are [1] to characterise the longitudinal trends of patient-measured FVC and PROM in a cohort of patients with IPF [2] to determine the correlation (if any) between patient-measured FVC and PROMs with clinic-observed measurements and [3] to assess if longitudinal trends in patient-measured FVC are predictive of clinical health outcomes in IPF. An additional purpose is to assess the acceptability and utility of the patientMpower app in helping IPF patients and their healthcare professional caregivers manage their condition. This app has been specially developed for patients with lung fibrosis and is owned by patientMpower Ltd., Dublin, Ireland. The app is downloaded to the patient's mobile phone/tablet device. Patients can record symptoms (e.g. dyspnea), activity (steps/day) and lung function (FVC) via a Bluetooth-connected hand-held spirometer. The app can also be used to remind patients to take their medicines. The app includes a PROM to capture impact of IPF on daily life (once/week).

This planned observation period is sixteen weeks. No additional clinic visits are required (compared with usual care). Only patients with a confirmed diagnosis of IPF who provide written informed consent will participate.

At a usual care visit to the IPF clinic at the study centre, the research team will discuss the study with the patient (face-to-face) and seek written informed consent. The study starts at this visit (baseline). The IPF clinic will record the usual measurements which would be done at a routine visit to assess IPF. These will include FVC, assessment of dyspnea (modified Medical Research Council score) and PROM.

After written informed consent, patientMpower Ltd. will send an information pack via e-mail and a Medical International Research Spirobank Smart spirometer to the patient. Technical support on installation of the app and spirometer will be provided by patientMpower Ltd. The patient will use the patientMpower app to record lung function, breathlessness, adherence to medication and symptoms every day at home until their next visit to the IPF clinic. Every week, patients will be reminded to record the impact of IPF on daily life PROM on the app. There will be no changes to the patient's usual care (e.g. prescribed medicines or exercises) during the study.

After about sixteen weeks, patients will return to the IPF clinic for routine assessment of their IPF. The clinic will record all of the usual measurements as at baseline. Patients and healthcare professionals will provide their opinion on the utility and acceptability of the patientMpower app. The study is concluded at this visit. However, patients can continue to use the patientMpower app and spirometer if they wish.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of idiopathic pulmonary fibrosis
* daily unrestricted access to smartphone/tablet device
* has an email address
* has home broadband or mobile data package
* demonstrates understanding of correct use of spirometer and patientMpower app
* able and willing to perform spirometry at home and record information on patientMpower app daily
* gives written informed consent

Exclusion Criteria:

* significant confusion or any concomitant medical condition which would limit teh ability of the patient to record symptoms or use a home spirometer regularly
* new prescription of antifibrotic therapy for IPF (e.g. pirfenidone, nintedanib) within four weeks of baseline visit
* recent exacerbation of IPF or other clinically significant change in patient's medical condition in the four weeks before the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic pulmonary fibrosis attending a specialist outpatient interstitial lung disease clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Respiratory Medicine, Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated: All patients who gave informed consent, downloaded the patientMpower application and used the patientMpower application with a MIR Spirobank Smart spirometer at least once. All patients received usual care throughout (i.e. no changes to care mandated by protocol.)
Period: Overall Study
Arm/Group | Treated
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Treated: All patients who gave informed consent, downloaded the patientMpower application and used the patientMpower application with a MIR Spirobank Smart spirometer at least once.
Arm/Group | Treated
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 20
In-clinic Forced Vital Capacity (absolute) [Mean (Standard Deviation); unit: Litres] | 3.30 (0.74)
In-clinic Forced Vital Capacity (percent predicted) [Mean (Standard Deviation); unit: percent predicted] | 92 (17)

OUTCOME MEASURES:

1. Primary Outcome: Patient-measured Spirometry Trend Over Time
Description: Mean patient-measured Forced Vital Capacity (FVC) in last seven days - FVC in first seven days after baseline
Time Frame: First 7 days at baseline and last 7 days in study up to 116 days
Measure: Mean (Standard Deviation); unit: litre
Arm/Group | Treated
Number analyzed (Participants) | 20
litre | -0.035 (0.490)

2. Primary Outcome: Correlation Between Patient-measured and Clinic-measured Spirometry at Baseline
Description: Bootstrap distribution of correlations analysis of patient-measured versus clinic-measured Forced Vital Capacity (FVC) at baseline calculated as follows. Means of first 7 days of patient-recorded FVC after baseline were calculated. (Patients without a single spirometry value in the 7-day window were excluded). Correlation between in-clinic FVC and patient-recorded FVC was calculated by randomly sampling from the data and calculating the Pearson correlation coefficient. This was repeated 1000 times, giving an empirical distribution for correlation (known as bootstrapping). The mean of this distribution is the inferred correlation.
Time Frame: First 7 days after baseline
Population: Patients in treated dataset for whom data were available in 7 days after baseline
Measure: Mean (Standard Deviation); unit: Distribution of correlation coefficient
Arm/Group | Treated
Number analyzed (Participants) | 9
Distribution of correlation coefficient | 0.72 (0.02)

3. Primary Outcome: Correlation Between Patient-measured and Clinic-measured Spirometry at End of Study
Description: Bootstrap distribution of correlations analysis of patient-measured versus clinic-measured Forced Vital Capacity (FVC) at end of study calculated as follows: Means of last 7 days of patient-recorded FVC after baseline were calculated. (Patients without a single spirometry value in the 7-day window were excluded). Correlation between in-clinic FVC and patient-recorded FVC was calculated by randomly sampling from the data and calculating the Pearson correlation coefficient. This was repeated 1000 times, giving an empirical distribution for correlation (known as bootstrapping). The mean of this distribution is the inferred correlation.
Time Frame: Last 7 days before end-of-study clinic visit
Population: Patients in treated dataset for whom data were available in the 7 days before end of study
Measure: Mean (Standard Deviation); unit: Distribution of correlation coefficient
Arm/Group | Treated
Number analyzed (Participants) | 13
Distribution of correlation coefficient | 0.77 (0.01)

4. Secondary Outcome: In-clinic Patient Reported Outcome Measure at Start
Description: Idiopathic Pulmonary Fibrosis Patient Reported Outcome Measure. Combined score from 4 domains (psychological & physical impact of breathlessness, psychological well-being, fatigue). Values range: 1-4. Higher scores indicate worse outcome. Reported by patient at clinic.
Time Frame: Baseline
Population: Patients reporting outcomes at beginning
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated
Number analyzed (Participants) | 20
score on a scale | 1.76 (0.76)

5. Secondary Outcome: In-clinic Patient Reported Outcome Measure at End
Description: as for outcome 4
Time Frame: End-of-study (116 days)
Population: Patients reporting outcomes at end
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated
Number analyzed (Participants) | 17
score on a scale | 1.78 (0.83)

6. Secondary Outcome: Patient-reported Patient Reported Outcome Measure at Start
Description: Idiopathic Pulmonary Fibrosis Patient Reported Outcome Measure. Combined score from 4 domains (psychological & physical impact of breathlessness, psychological well-being, fatigue). Values range: 1-4. Higher scores indicate worse outcome. Reported by patient at home.
Time Frame: Baseline
Population: Patients reporting outcome measure at home (not available for all subjects entered)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated
Number analyzed (Participants) | 10
score on a scale | 1.60 (0.60)

7. Secondary Outcome: Patient-reported Patient Reported Outcome Measure at End
Description: Idiopathic Pulmonary Fibrosis Patient Reported Outcome Measure; psychological & physical impact of breathlessness, psychological well-being, fatigue domains, values range 1-4, higher scores worse outcome. Reported by patients at home.
Time Frame: End-of-study (116 days)
Population: Patients reporting outcome measure at home (not available for all subjects entered)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treated
Number analyzed (Participants) | 9
score on a scale | 1.79 (0.93)

8. Secondary Outcome: In-clinic Dyspnea Score at Start
Description: modified Medical Research Council dyspnea score (range 0-4; worst dyspnea = 4)
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treated
Number analyzed (Participants) | 20
score on a scale | 2 [1.75 to 2.25]

9. Secondary Outcome: In-clinic Dyspnea Score at End
Description: modified Medical Research Council dyspnea score (range 0-4; worst dyspnea = 4)
Time Frame: 116 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treated
Number analyzed (Participants) | 16
score on a scale | 2 [1 to 2]

10. Secondary Outcome: Patient Opinion: Instructions Understandable?
Description: Number of subjects responding "strongly agree" or "agree" shown. 4 possible responses: strongly agree/agree/disagree/strongly disagree;
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 10

11. Secondary Outcome: Patient Opinion: Helped me Take Correct Dose of Medicines?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 9

12. Secondary Outcome: Patient Opinion: Helped me Achieve Exercise Goal?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 9

13. Secondary Outcome: Patient Opinion: Helped me Walk Further?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 6

14. Secondary Outcome: Patient Opinion: Using Application Gave me More Confidence?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 8

15. Secondary Outcome: Patient Opinion: Useful to Measure Impact of Pulmonary Fibrosis on Daily Life?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 9

16. Secondary Outcome: Patient Opinion: I Liked Using the Application?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 10

17. Secondary Outcome: Patient Opinion: the Application Was Easy to Use?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 9
Participants | 9

18. Secondary Outcome: Patient Opinion: it Was Irritating to Use the Application?
Description: as for outcome 10
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 1

19. Secondary Outcome: Patient Opinion: Was the Effect of Application on Impact on Daily Life Positive?
Description: Number of subjects responding "yes". 2 possible responses: yes/no
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 9

20. Secondary Outcome: Patient Opinion: I Want to Continue Using the Application?
Description: Number of subjects responding "yes". 2 possible responses: yes/no
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 9

21. Secondary Outcome: Patient Opinion: I Would Recommend the Application to Others?
Description: Number of subjects responding "yes". 2 possible responses: yes/no
Time Frame: 116 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treated
Number analyzed (Participants) | 10
Participants | 9

ADVERSE EVENTS:
Time Frame: 128 +/- 34 days (mean +/- standard deviation)
Arm/Group | Treated
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treated (N=20)
Sore throat (Gastrointestinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
dizziness (General disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
loss of appetite (Gastrointestinal disorders) | 1
headache (General disorders) | 1
anxiety (Psychiatric disorders) | 1
Exacerbation idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT03744598/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT03744598/SAP_001.pdf